CLINICAL TRIAL: NCT06186531
Title: PhytoSERM for Menopausal Hot Flashes and Sustained Brain Health: A Double-Blind, Randomized, Placebo-Controlled Phase 2 Clinical Trial
Brief Title: PhytoSERM for Menopausal Hot Flashes and Sustained Brain Health
Acronym: HF-Relief
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuTherapeutics (Industry)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phyto-HF-2022-01
Record Dates: First submitted 2023-11-30; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Menopause; Hot Flashes
Keywords: Phytoestrogen supplement; Menopause; Hot flashes; Cognition
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, parallel group design with open-label extension.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PhytoSERM (Experimental): Active intervention group
  Interventions: Dietary Supplement: PhytoSERM
- Placebo group (Placebo Comparator): Control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: PhytoSERM — PhytoSERM, a formulated dietary supplement, will be an ovalized tablet measuring 8.51 mm x 15.49 mm. Each pill will contain a white PEG coating and an equal mixture of, daidzein, genistein, and S-equol.
  Arms: PhytoSERM
Drug: Placebo — Placebo product is of identical shape, size and color with a white PEG coating but without S-equol, daidzein and genistein.
  Arms: Placebo group

SUMMARY:
This is a proof-of-concept phase 2 clinical trial to investigate the effect of the phytoestrogenic supplement PhytoSERM on vasomotor symptoms and other symptoms associated with the menopausal transition, and on blood-based biomarkers in peri- and postmenopausal women.

After the screening period, participants will be randomized to PhytoSERM 50 mg pills (administered orally, once per day) or matching placebo, 1:1 allocation, for a period of 12 weeks. After 12 weeks, all participants in the placebo group will be crossed-over to receive PhytoSERM pills for the remainder of the study (open-label phase).

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled, parallel designed, proof-of-concept phase 2 clinical trial to determine effect of PhytoSERM on vasomotor symptoms and other symptoms associated with the menopausal transition. PhytoSERM or placebo pills will be administered orally once a day over 24 weeks. Safety and tolerability will also be assessed over the duration of the study.

A total of 132 peri- or postmenopausal women aged 45-60 years and who are experiencing hot flashes will be enrolled in this trial. To determine eligibility, all participants will undergo cognitive assessment, physical assessment, ECG, clinical/safety laboratory assessment, and interviews. After a 2-week screening period, participants will be randomized to study intervention (PhytoSERM 50mg administered orally, once per day) or matching placebo, in a 1:1 allocation. After 12 weeks, participants in the placebo group will be crossed-over to PhytoSERM 50 mg for the remaining 12 weeks (open-label extension period). Hot flashes will be measured both objectively and subjectively. Objective data will be skin conductance levels collected via a wearable device that enables real-time physiological data acquisition, including activity and sleep data. Study participants will be asked to complete a total of 8 study visits. Study visits will occur at 4-week intervals after the baseline, except for visits # 6 and 7 (open-label period) which will occur at 6-week intervals after visit # 5 (final outcomes assessments visit). Visits 1, 2, 5 and 7 will last approximately 2-4 hours; visits 3, 4, 6 and 8 will last approximately 45 minutes.

All participants will be enrolled at a single site, at the University of Arizona (UA) Clinical & Translational Sciences Research Center (CATS).

ELIGIBILITY:
Inclusion Criteria:

* Peri- or postmenopausal women, defined by any of the following:

  1. Last menstrual period (LMP) completed ≥ 60 days and ≤ 8 years, per the Stages of Reproductive Aging Workshop (STRAW) criteria.
  2. Post-hysterectomy or endometrial ablation ≥ 3 months and supported by FSH levels.
* Age 45-60 years.
* Presence of hot flashes ≥ 7 per day.
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be not clinically significant by the investigator.
* Mammogram within normal limits in the past 2 years: Breast Imaging Reporting and Data System (BI-RADS) category 1-2 or 3 with findings stable for 3 years.
* No medical contraindications to study participation.
* Stable medications for 4 weeks prior to the baseline visits.
* Ability to take oral medication and be willing to adhere to the PhytoSERM regimen.
* For females of reproductive potential: Negative pregnancy test and use of highly effective contraception by male partner for at least 1 month prior to screening and agreement to use such a method during study participation.

Exclusion Criteria:

* Use of isoflavone containing supplements.
* Known allergies to isoflavones or soy-based products.
* Montreal Cognitive Assessment total score < 22.
* Pregnancy
* Use of estrogen or progestin compounds within 8 weeks of baseline.
* Use of investigational agent within 12 weeks of baseline.
* Concurrent neurologic, systemic, or psychiatric disease that would influence cognition or ability to provide informed consent and to participate.
* Known or suspected estrogen-dependent neoplasia (breast, ovarian and uterine cancers), active neoplastic disease, history of breast cancer, and endometrial hyperplasia.
* History within the last 5 years of any other primary or recurrent malignant disease, with the exception of resected cutaneous squamous cell carcinoma in situ, and basal cell carcinoma.
* History of epilepsy, focal brain lesion, head injury with loss of consciousness or DSM IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol, or substance abuse.
* Thrombophlebitis, thrombosis, thromboembolic disorders, myocardial infarction, ischemic heart disease, cerebrovascular accident, stroke, TIA.
* Current use of tobacco or a history of alcohol abuse.
* Use of anticoagulants.
* Chronic use of most benzodiazepines
* Use of drugs, herbs, or dietary supplements to treat menopausal or cognitive symptoms less than 8 weeks prior to baseline (e.g., SSRIs, rhubarb, red clover, licorice, kudzu, black cohosh, ginseng or other similar roots, etc.)
* Evidence of any significant clinical disorder or laboratory finding, including clinically significant or unstable hematologic, hepatic, cardiovascular, pulmonary, gastrointestinal, endocrine, metabolic, renal, or other systemic disease or laboratory abnormality.
* Known allergy to soy-derived products/ proteins or branded over the counter products; hypersensitivity to estrogens or progestins.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Peri and postmenopausal women
Enrollment: 132 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Hot Flash Composite score | Daily from baseline to week 24
  Composite score comprised by hot flash frequency and severity (sum of weekly hot flashes weighted by severity: mild, moderate, severe). Higher score indicates a bad outcome. No minimum or maximum values.

SECONDARY OUTCOMES:
Trail Making Test score | Baseline, week 4, 8, 12 and 24.
  Test that involves visual scanning and working memory. Score is the amount of seconds taken to complete the test; the greater the time the worse the score.
NIH Toolbox List Sorting Working Memory Test score | Baseline, week 4, 8, 12 and 24.
  An assessment of working memory administered on an iPad. Scores range from 0 to 26, with higher being better.
NIH Toolbox Picture Sequence Memory Test | Baseline, week 4, 8, 12 and 24.
  An assessment of episodic memory administered on an iPad. The participants are asked to recall the sequence of pictures demonstrated over two learning trials; sequence length varies from 6-18 pictures. Participants are given credit for each adjacent pair of pictures they correctly place up to the maximum value for the sequence, which is one less than the sequence length. Range is 0-17.
NIH Toolbox Auditory Verbal Learning Test | Baseline, week 4, 8, 12 and 24.
  An assessment of immediate memory and verbal learning administered on an iPad.Possible range is 0-45 words, with higher scores representing better performance.
NIH Toolbox Oral Symbol Digit Test | Baseline, week 4, 8, 12 and 24.
  An assessment of processing speed administered on an iPad. Scored as the number of items answered correctly in 120 seconds (possible range is 0-144).
Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 4, 8, 12, 18, 24 and 28.
  Instrument used to measure the quality patterns of sleep in the older adult. A global sum of "5" or greater indicates a "poor" sleeper.
Menopause Rating Scale score | At screening, weeks 12, 24 and 28.
  A a health-related quality of life scale measuring the impact of menopausal symptoms. The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints).
Bone Mineral Density (BMD) | Baseline, week 12 and 24
  BMD in g/cm2 will be measured with a Dual-energy X-ray absorptiometry (DXA) scan. Expected range is 0.5-1.5 g/cm2, with higher being better.
Bone Mineral Content (BMC) | Baseline, week 12 and 24
  BMC in grams will be measured with a Dual-energy X-ray absorptiometry (DXA) scan. Expected range is 2,000 - 3,500 g, with higher being better.
Body Mass Index (BMI) | Baseline, week 12 and 24
  BMI will be measured with a Dual-energy X-ray absorptiometry (DXA) scan. Range is 10-45.
Total Fat Mass (TFM) | Baseline, week 12 and 24
  TFM in grams will be measured with a Dual-energy X-ray absorptiometry (DXA) scan.
Total Lean Mass (TLM) | Baseline, week 12 and 24
  TLM in grams will be measured with a Dual-energy X-ray absorptiometry (DXA) scan.

OTHER OUTCOMES:
Digital hot flash frequency | Daily from baseline to week 28.
  Skin conductance levels measured via electrodermal activity (EDA) sensors will be used as an objective physiological measure of hot flashes.
Follicle-Stimulating Hormone (FSH) levels | Baseline, weeks 12 and 24
  Reproductive hormone / menopause biomarker
Estrodiol levels | Baseline, weeks 12 and 24
  Reproductive hormone / menopause biomarker
Cholesterol levels | Baseline, weeks 12 and 24
  Metabolic biomarker
Trigliceryde levels | Baseline, weeks 12 and 24
  Metabolic biomarker
HbA1C levels | Baseline, weeks 12 and 24
  Metabolic biomarker
Aß40:Aß42 ratio | Baseline, weeks 12 and 24
  Alzheimer's biomarker
Glial fibrillary acidic protein (GFAP) levels | Baseline, weeks 12 and 24
  Neuroinflammation biomarker
Neurofilament Light (NfL) levels | Baseline, weeks 12 and 24
  Neurodegeneration biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Fei Yin, PhD, Principal Investigator — University of Arizona; Gerson D Hernandez, MD, MPH, Study Director — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States